CLINICAL TRIAL: NCT03025789
Title: An Open-label Study Assessing Effectiveness, Safety and Compliance With Fexinidazole in Patients With Human African Trypanosomiasis Due to T.b. Gambiense at Any Stage
Brief Title: Fexinidazole in Human African Trypanosomiasis Due to T.b. Gambiense at Any Stage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-FEX-09-HAT
Record Dates: First submitted 2016-11-11; First posted 2017-01-20 (Estimated); Results first posted 2024-06-07 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Trypanosomiasis, African; Sleeping Sickness; Trypanosomiasis; Gambian
Keywords: T.b gambiense; HAT; outpatients
MeSH Terms: conditions — Trypanosomiasis, African; Trypanosomiasis | interventions — fexinidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inpatients (Experimental): Participants received fexinidazole orally for 10 days as inpatients (at the hospital)
  Interventions: Drug: Fexinidazole
- Outpatients (Experimental): Participants received fexinidazole orally for 10 days as outpatients (at home)
  Interventions: Drug: Fexinidazole

INTERVENTIONS:
Drug: Fexinidazole — Tablets of 600 mg; Participants with a weight between 20 and 34 kg received 1200 mg (2 tablets) for 4 days, then 600 mg (1 tablet) for 6 days (with food); Participants with a weight of 35 kg and above received 1800 mg (3 tablets) for 4 days, then 1200 mg (2 tablets) for 6 days (with food)

SUMMARY:
This study evaluates the effectiveness of fexinidazole administered to patients with human African trypanosomiasis due to T. b. gambiense (g-HAT) at all stages of the disease. The aim of the present study is to provide additional information on the effectiveness and safety of fexinidazole and to assess its use under conditions as close as possible to those in real life, both in patients treated on an out-patient basis and in the hospital setting, depending on clinical status.

Participants will receive fexinidazole oral treatment for 10 days. Regular blood draws and lumbar punctures will be performed over 18 months to confirm the cure of the disease. Other assessments will include the recording of adverse events, signs and symptoms of the disease, laboratory tests, vital signs, electrocardiograms. Treatment compliance, feasibility, and packaging acceptability will be thoroughly assessed in the participants receiving treatment at home. Those participants will complete questionnaires to check that instructions for fexinidazole administration are clear enough and followed correctly.

DETAILED DESCRIPTION:
See attached protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, including breastfeeding or pregnant women in the second or third trimester.
* ≥ 6 years of age.
* ≥ 20 kg body weight.
* Signed Informed Consent Form and Assent Form for patients less than 18 years of age
* Trypanosomes detected in any body fluid.
* Physically able to ingest at least one solid meal per day.
* Able to take oral medication.
* Karnofsky Performance Status > 40%.
* Able to comply with the schedule of follow-up visits and with the study constraints.
* Easily reachable during the out-patient follow-up period.
* Willing to undergo lumbar punctures.

Exclusion Criteria:

* Active clinically relevant medical conditions other than HAT that, in the Investigator's opinion, could jeopardize patient safety or interfere with participation in the study, including but not limited to significant liver or cardiovascular diseases, human immunodeficiency virus (HIV) infection, central nervous system (CNS) trauma or seizure disorders, coma or altered consciousness not related to HAT.
* Severe renal or hepatic impairment defined as:

elevated creatinine at > 3 times the upper limit of normal (ULN); elevated alanine aminotranferase (ALT), aspartate aminotransferase (AST), or bilirubin at > 3 ULN

* Severely deteriorated general condition, such as cardiovascular shock, respiratory distress or terminal illness.
* Any condition (except symptoms of HAT) that compromises ability to communicate with the Investigator as required for completion of the study.
* Any contraindication to imidazole products (known hypersensitivity to imidazoles).
* Treatment for HAT within 2 years prior to inclusion.
* Prior enrolment in the study or prior intake of fexinidazole.
* Foreseeable difficulty in complying with the schedule of follow-up visits (migrants, refugees, itinerant traders, etc.).

Temporary Non-inclusion Criteria:

* Recovery period after antimalarial treatment and/or treatment of helminthiasis (at least 3 days).
* Uncontrolled diabetes or hypertension or any patients requiring clinical stabilization; wait until appropriate treatment to control the disease has been initiated.
* First trimester of pregnancy.
* Traumatic lumbar puncture at Screening i.e. red blood cells visible in cerebrospinal fluid (CSF); wait for 48 hours before repeating lumbar puncture.

Eligibility Criteria for Out-patient Treatment

* Accepting to be treated on an out-patient basis;
* Karnofsky Performance Status > 50%;
* Good understanding of the method of administration of fexinidazole by the patient and/or caregiver* (checked using a questionnaire at the time of dispensing fexinidazole);
* Residing close to the investigational center, i.e. approximately one hour by road and/or boat, during the treatment period**;
* Easily reachable during the treatment period;
* No medical or psychiatric contraindications for treatment as out-patient;
* No pregnancy or breastfeeding;
* No neurological symptoms.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Kande Betu Kumeso, MD, Principal Investigator — Ministry of Health, Kinshasa, The Democratic Republic of the Congo; Mamadou Camara, PhD, Principal Investigator — National HAT Control Programme, Conakry, Guinea; Médard Ilunga Wa Kyhi, MD, Principal Investigator — National HAT Control Programme, Kinshasa, The Democratic Republic of the Congo; Digas Ngolo Tete, MPH, Principal Investigator — National HAT Control Programme, Kinshasa, The Democratic Republic of the Congo
Locations (8):
- Democratic Republic of the Congo (7):
  - Dipumba Hospital, Mbuji-Mayi, Kasaï Oriental Province
  - Bagata Hospital, Bagata, Kwilu
  - Bandundu Hospital, Bandundu Province, Kwilu
  - Masi Manimba Hospital, Masi-Manimba, Kwilu
  - Nkara Secondary Hospital, Nkara, Kwilu
  - Mushie Hospital, Mushie, Maï Ndombe Province
  - Roi Baudouin Hospital, Kinshasa
- Dubreka Hospital, Dubréka, Guinea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO. Human African trypanosomiasis: update of the methodological framework for clinical trials: report of the first meeting of the Development of New Tools subgroup, Geneva, 24 September 2014. World Health Organization 2015. WHO/HTM/NTD/IDM/2015.5
- [Derived] Kumeso VKB, Perdrieu C, Menetrey C, Kyhi MIW, Tete DN, Camara M, Tampwo J, Kavunga P, Camara ML, Kourouma A, Mindele WK, Masa FA, Mahenzi H, Makaya J, Malu TM, Mandula G, Nzambi DMM, Ntoya SL, Reymondier A, Kalonji WM, Scherrer B, Mordt OV. Effectiveness and safety of fexinidazole for gambiense human African trypanosomiasis and exploration of adherence in outpatients: a phase 3b, prospective, open-label, non-randomised, cohort study. Lancet Glob Health. 2025 May;13(5):e900-e909. doi: 10.1016/S2214-109X(24)00526-6. PMID 40288399

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 8 centers in the Democratic Republic of Congo and 1 center in Guinea. 200 participants were screened and signed informed consent. 3 patients had no trypanosomes in their blood and were not included since g-HAT positivity could not be confirmed. Of the 197 screened HAT-positive participants, 174 were included and treated, and 23 were not included, mainly due to inclusion/exclusion criteria not met. Participants were enrolled between 10 November 2016 and 10 August 2019.
Pre-assignment Details: The pre-treatment period of up to 15 days included screening and treatment of concurrent malaria/soil-transmitted helminthiasis. At the end of this period, all participants (regardless of g-HAT stage and treatment setting) were treated with fexinidazole.
Period: Overall Study
Arm/Group | Inpatients | Outpatients
Started | 136 | 38
Completed | 129 | 35
Not Completed | 7 | 3
Not completed — Lack of Efficacy | 6 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (mITT) population included all participants who received at least one tablet of fexinidazole.
Groups:
- Total: Total of all reporting groups
Arm/Group | Inpatients | Outpatients | Total
Number analyzed (Participants) | 136 | 38 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (15.5) | 27.9 (18.0) | 26.4 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 18 | 96
  Male | 58 | 20 | 78
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Sub-Saharan African | 136 | 38 | 174
Region of Enrollment [Count of Participants; unit: Participants]
  Guinea | 26 | 6 | 32
  Congo, The Democratic Republic of the | 110 | 32 | 142
g-HAT stage: Stage 1/intermediate, Stage 2 [Count of Participants; unit: Participants] — Patients with trypanosomes in the cerebrospinal fluid (CSF) were classified as "stage 2". Patients without trypanosomes in the CSF were classified as "stage 1" if white blood cells (WBC) count in CSF ≤5 /µL, "intermediate stage" if WBC in CFS ≥6 and ≤20 /µL, or "stage 2" if WBC in CSF >20 /µL.
  Participants
    Stage 1/intermediate | 53 | 17 | 70
    Stage 2 | 83 | 21 | 104
White blood cell (WBC) in cerebrospinal fluid (CSF) [Count of Participants; unit: Participants]
  100 cells/µL or lower | 80 | 20 | 100
  Higher than 100 cells/µL | 56 | 18 | 74

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Whose Treatment Outcome at Month 18 is a Success
Description: Treatment outcome at Month 18 is categorized as success or failure. Success is defined as a cure, according to the criteria adapted from the World Health Organization (WHO) update of the methodological framework for clinical trials in Sept 2014 (WHO/HTM/NTD/IDM/2015.5). Failure is defined as a relapse, probable relapse, death, use of rescue medication, loss to follow-up, refusal of all post-treatment lumbar puncture, and, in the absence of lumbar puncture at the Month 18 visit, an unfavorable outcome earlier than Month 18, or signs and symptoms evoking a relapse at Month 18. Success rate at Month 18 is defined as the percentage of participants (regardless of g-HAT stage) whose treatment outcome is a success at Month 18. An estimate of the success rate at Month 18 and the 95% exact Clopper-Pearson confidence interval (CI) of the estimate are provided.
Time Frame: Between the first intake of fexinidazole (Day 1) and the end of the follow-up period (18 months)
Population: This population includes all patients in the mITT population (i.e. who received at least one table of fexinidazole), regardless of treatment setting (inpatients and outpatients). The efficacy of fexinidazole was not meant to be studied in inpatients and outpatients separately.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Treated Patients, Regardless of Treatment Setting: Participants were to receive fexinidazole orally for 10 days, either as outpatients (at home) or as inpatients (at the hospital)
Arm/Group | All Treated Patients, Regardless of Treatment Setting
Number analyzed (Participants) | 174
percentage of participants | 93.1 [88.3 to 96.4]

2. Secondary Outcome: Percentage of Participants Whose Treatment Outcome at Month 12 is a Success
Description: Treatment outcome at Month 12 is categorized as success or failure. Success is defined as a cure, according to the criteria adapted from the World Health Organization (WHO) update of the methodological framework for clinical trials in Sept 2014 (WHO/HTM/NTD/IDM/2015.5). Failure is defined as a relapse, probable relapse, death, use of rescue medication, loss to follow-up, refusal of all post-treatment lumbar puncture, and, in the absence of lumbar puncture at the Month 12 visit, an unfavorable outcome earlier than Month 12, or signs and symptoms evoking a relapse at Month 12 (data collected at Month 18 are considered, if available). Success rate at Month 12 is defined as the percentage of participants (regardless of g-HAT stage) whose treatment outcome is a success at Month 12. An estimate of the success rate at Month 12 and the 95% exact Clopper-Pearson confidence interval (CI) of the estimate are provided.
Time Frame: Between the first intake of fexinidazole (Day 1) and the end of the follow-up period (18 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Treated Patients, Regardless of Treatment Setting
Number analyzed (Participants) | 174
percentage of participants | 94.3 [89.7 to 97.2]

3. Secondary Outcome: Number of Participants With Any Grade ≥ 3 Treatment-emergent Adverse Events (AEs) Including Laboratory and Hematological Abnormalities (if Considered Clinically Significant)
Description: AE severity is graded according to the National Cancer Institute (NCI) Common Toxicity Criteria for AEs (CTCAE), Version 4.03 and, for certain laboratory parameters, modified CTCAE is used. Grade ≥3 AEs include the following events: Grade 3 events (severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living), Grade 4 events (life-threatening consequences; urgent intervention indicated), and Grade 5 events (death related to AE).
  The observation period extends from the first intake of fexinidazole (Day 1) until the end-of-hospitalization visit (between Day 13 and Day 18) for inpatients and until the end-of-treatment visit (on Day 11) for outpatients.
Time Frame: Between the first intake of fexinidazole (Day 1) and the end of the observation period, or the end of the follow-up period (18 months) for non-serious AEs assessed as related to fexinidazole
Population: The mITT population included all participants who received at least one table of fexinidazole.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatients | Outpatients
Number analyzed (Participants) | 136 | 38
Participants | 10 | 4

4. Secondary Outcome: Number of Participants With Any Treatment-emergent Serious Adverse Event (SAE)
Description: An SAE was defined as any AE that: resulted in death; was life-threatening; required inpatient hospitalisation or prolongation of existing hospitalisation; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; was an important medical event that was not immediately life-threatening or did not result in death, but that jeopardised the patient's safety or required an intervention to prevent one of the outcomes above. Patients treated on an outpatient basis who required hospitalisation, for whatever reason, underwent the same procedures as patients initially treated in hospital, up to the end of the hospitalisation period. During this period, and up to Day 13 or Day 18, the reasons for hospitalisation were not to be considered to be SAEs solely based on the criterion of hospitalisation, but could be considered to be SAEs based on other criteria.
Time Frame: Between the first intake of fexinidazole (Day 1) and the end of the follow-up period (18 months)
Population: The mITT population included all participants who received at least one table of fexinidazole.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatients | Outpatients
Number analyzed (Participants) | 136 | 38
Participants | 10 | 4

5. Secondary Outcome: Number of Participants With Any Temporary or Permanent Treatment Discontinuation (Inpatient or Outpatient) for Reasons Related to Safety
Description: Number of patients who prematurely discontinued treatment (temporarily or permanently) for reasons related to safety (including overdose).
Time Frame: Between the first intake (Day 1) and last intake of fexinidazole (Day 10, or Day 11 if re-administration occurred)
Population: The mITT population included all participants who received at least one table of fexinidazole.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatients | Outpatients
Number analyzed (Participants) | 136 | 38
Participants | 4 | 0

6. Secondary Outcome: Number of Participants With Any Hospitalization for Reasons Related to Safety (Outpatients Only)
Description: Number of outpatients who are hospitalized for reasons related to safety (including overdose). An outpatient is considered as "hospitalized for reasons related to safety" if he/she is initially planned to be treated as an outpatient but experiences an AE during the treatment period (Day 1 to Day 10) and is hospitalized during the treatment period.
Time Frame: Between the first intake (Day 1) and last intake of fexinidazole (Day 10, or Day 11 if re-administration occurred)
Population: All outpatients included in the mITT population (i.e. who received at least one table of fexinidazole). This outcome measure is only applicable to outpatients to investigate the proportion of outpatients who had to be hospitalized during treatment due to safety.
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatients
Number analyzed (Participants) | 38
Participants | 2

7. Secondary Outcome: Number of Participants With Any Permanent Treatment Discontinuation (Inpatient or Outpatient) for Reasons Related to Safety
Description: Number of patients who prematurely discontinued treatment permanently for reasons related to safety (including overdose).
Time Frame: Between the first intake (Day 1) and last intake of fexinidazole (Day 10, or Day 11 if re-administration occurred)
Population: The mITT population included all participants who received at least one table of fexinidazole.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatients | Outpatients
Number analyzed (Participants) | 136 | 38
Participants | 1 | 0

8. Secondary Outcome: Number of Outpatients Who Were Compliant With the Full Course of the 10-day Treatment
Description: Number of outpatients who completed the full course of the 10-day treatment. Full completion can be either completing the 10-day treatment in the outpatient setting, or starting treatment as an outpatient but finishing treatment at the hospital, for those who have to be hospitalized (for any reason). At Day 11, the participant and/or caregiver have to present the treatment packaging they received at study inclusion, and the investigator has to record if the treatment calendar was fully completed or not.
Time Frame: Between the first intake (Day 1) and last intake of fexinidazole (Day 10, or Day 11 if re-administration occurred)
Population: All outpatients included in the mITT population (i.e. participants who received at least one tablet of fexinidazole).
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatients
Number analyzed (Participants) | 38
Participants | 38

9. Secondary Outcome: Number of Outpatients Who Were Compliant With the 10-day Treatment Posology, Including Taking the Correct Number of Tablets During the 2 Phases of Treatment and Taking Tablets All at Once Every Day, With Food and Without Any Interruption of Treatment
Description: Number of patients whose response to the question "How did you take your treatment?" is correct, as determined by the study personnel leading the compliance interview at Day 11 (end-of-treatment visit).
  The expected answer for participants weighing 35 kg or more is: 2 phases. Day 1 to 4 = 3 tablets. Day 5 to 10 = 2 tablets. Tablets to be taken all at once during a meal.
  The expected answer for participants weighing less than 35 kg is: 2 phases. Day 1 to 4 = 2 tablets. Day 5 to 10 = 1 tablet. Tablets to be taken all at once during a meal.
  The answer is considered correct if the 4 key messages have been understood (treatment period composed of 2 phases, each with a different number of tablets to be taken; treatment to be taken for 10 days without interruption; tablets to be taken all at once every day; treatment to be taken during a meal)
Time Frame: End-of-treatment visit (Day 11)
Population: Three of the 38 outpatients included in the mITT population were hospitalized and completed treatment at the hospital. As a consequence, they did not fill out the compliance questionnaire designed for outpatients after treatment. Therefore, the total number of patients analyzed was 35 outpatients.
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatients
Number analyzed (Participants) | 35
Participants | 35

10. Secondary Outcome: Feasibility of Self-management of Treatment Intake in Outpatients: Occurrence of Temporary Treatment Discontinuation
Description: The occurrence of temporary treatment discontinuation is recorded at Day 11 (end-of-treatment visit) in the case report form by the study personnel (Section on feasibility, question "Was the treatment temporarily discontinued?). Occurrence is presented as the number of outpatients who temporarily discontinued their treatment.
Time Frame: End-of-treatment visit (Day 11)
Population: All outpatients included in the mITT population (i.e. who received at least one table of fexinidazole).
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatients
Number analyzed (Participants) | 38
Participants | 0

11. Secondary Outcome: Feasibility of Self-management of Treatment Intake in Outpatients: Occurrence of Permanent Treatment Discontinuation
Description: The occurrence of permanent treatment discontinuation is recorded at Day 11 (end-of-treatment visit) in the case report form by the study personnel (Section on feasibility, question "Was the treatment stopped permanently?). Occurrence is presented as the number of outpatients who prematurely (prior to Day 10) discontinued their treatment permanently.
Time Frame: End-of-treatment visit (Day 11)
Population: All outpatients included in the mITT population (i.e. who received at least one table of fexinidazole).
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatients
Number analyzed (Participants) | 38
Participants | 0

12. Secondary Outcome: Feasibility of Self-management of Treatment Intake in Outpatients: Delayed Treatment Start
Description: The occurrence of delayed treatment start is recorded at Day 11 (end-of-treatment visit) in the case report form by the study personnel (Section on feasibility, date of first administration [Day 1] minus date of dispensing [Day 0] > 1 day). The occurrence of delayed treatment start is presented as the number of outpatients who had their planned treatment start delayed by at least 1 day.
Time Frame: End-of-treatment visit (Day 11)
Population: All outpatients included in the mITT population (i.e. who received at least one table of fexinidazole).
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatients
Number analyzed (Participants) | 38
Participants | 0

13. Secondary Outcome: Feasibility of Self-management of Treatment Intake in Outpatients: Hospitalization During the Treatment Period Due to Non-compliance
Description: The occurrence of hospitalization is recorded at Day 11 (end-of-treatment visit) in the case report form by the study personnel (Section on feasibility, question "Did the patient finish his/her treatment in hospital?"), with "non-compliance" as the reason for hospitalization. Occurrence of hospitalization is presented as the number of outpatients who had to be hospitalized during the treatment period due to non-compliance.
Time Frame: End-of-treatment visit (Day 11)
Population: All outpatients included in the mITT population (i.e. who received at least one table of fexinidazole).
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatients
Number analyzed (Participants) | 38
Participants | 1

14. Secondary Outcome: Acceptability of Packaging in Outpatients: Full Understanding of Instructions Concerning Dosing Regimen
Description: Full understanding of the instructions concerning the dosing regimen of fexinidazole is assessed at Day 0 (day of treatment dispensing) by the study personnel. During the interview, the study personnel ask the participant and/or caregiver 8 questions about posology. To each of these 8 questions, the study personnel tick 'Yes' if the immediate answer is consistent with the expected answer. Full understanding of the instructions requires all 8 questions to be answered correctly. Full understanding is presented as the number of patients who correctly answered all 8 questions.
Time Frame: Before treatment (Day 0)
Population: All outpatients included in the mITT population (i.e. who received at least one table of fexinidazole).
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatients
Number analyzed (Participants) | 38
Participants | 30

15. Secondary Outcome: Acceptability of Packaging in Outpatients: Help Requested to Follow the Treatment
Description: Acceptability of packaging is assessed at Day 11 (end-of-treatment visit) by a questionnaire filled out by the participant and/or caregiver. The occurrence of help needed is presented as the number of outpatients who indicate at the end of treatment that they had to request help to follow the treatment (Section on acceptability, question "Did you have to request help to follow the treatment?").
Time Frame: End-of-treatment visit (Day 11)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatients
Number analyzed (Participants) | 35
Participants | 10

16. Secondary Outcome: Acceptability of Packaging in Outpatients: Instructions Found Helpful
Description: Acceptability of packaging is assessed at Day 11 (end-of-treatment visit) by a questionnaire filled out by the participant and/or caregiver. The number of patients who found the instructions helpful is recorded (Section on acceptability, question "Did you find the instruction sheet provided with the medication helpful / Did it help you to remember the important information?").
Time Frame: End-of-treatment visit (Day 11)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatients
Number analyzed (Participants) | 35
Participants | 35

17. Secondary Outcome: Whole Blood Concentration of Fexinidazole From Dry Blood Spot, Measured 24 Hours After the Last Dose of Fexinidazole
Description: Concentrations of fexinidazole is determined using a validated analytical method, in all patients with available PK data.
Time Frame: End-of-treatment visit (Day 11, 24 hours after last treatment administration)
Population: The PK population included all participants who received at least one table of fexinidazole and who had available PK data. The number of outpatients/inpatients in the PK analysis (36/138) differs from the main analysis (38/136) because 2 outpatients were hospitalized (on Day 3 and 5) and were considered as inpatients for the PK analysis (the outpatient hospitalized on Day 8 was considered as an outpatient for the PK analysis). Data were missing for 14 patients (10 inpatients and 4 outpatients).
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Inpatients | Outpatients
Number analyzed (Participants) | 128 | 32
µg/mL | 0.048 [0.01 to 0.27] | 0.054 [0.01 to 0.18]

18. Secondary Outcome: Whole Blood Concentration of Fexinidazole Metabolite M1 From Dry Blood Spot, Measured 24 Hours After the Last Dose of Fexinidazole
Description: Concentrations of fexinidazole metabolite M1 (fexinidazole sulfoxide) is determined using a validated analytical method, in all patients with available PK data.
Time Frame: End-of-treatment visit (Day 11, 24 hours after last treatment administration)
Population: The PK population included all participants who received at least one table of fexinidazole and who had available PK data. The number of outpatients/inpatients in the PK analysis (36/138) differs from the main analysis (38/136) because 2 outpatients were hospitalized (on Day 3 and 5) and were considered as inpatients for the PK analysis (the outpatient hospitalized on Day 8 was considered as an outpatient for the PK analysis). Data were missing for 1 patient (1 outpatient).
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Inpatients | Outpatients
Number analyzed (Participants) | 138 | 35
µg/mL | 1.928 [0.11 to 7.50] | 2.316 [0.13 to 4.41]

19. Secondary Outcome: Whole Blood Concentration of Fexinidazole Metabolite M2 From Dry Blood Spot, Measured 24 Hours After the Last Dose of Fexinidazole
Description: Concentrations of fexinidazole metabolite M2 (fexinidazole sulfone) is determined using a validated analytical method, in all patients with available PK data.
Time Frame: End-of-treatment visit (Day 11, 24 hours after last treatment administration)
Population: as for outcome 18
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Inpatients | Outpatients
Number analyzed (Participants) | 138 | 35
µg/mL | 11.014 [3.54 to 33.30] | 11.725 [2.55 to 35.86]

ADVERSE EVENTS:
Time Frame: Per protocol, non-serious adverse events (AEs) were recorded as follows: for inpatients, from the first intake of fexinidazole (Day 1) until the end-of-hospitalization Visit (Day 13-18) and in outpatients, from the first intake of fexinidazole (Day 1) until the end-of-treatment Visit (Day 11). Treatment-emergent serious AEs were collected from the first intake of fexinidazole (Day 1) until the end of the follow-up (Month 18). The population of analysis corresponds to the mITT population.
Description: Adverse events were classified as serious according to the standard definition. In addition, in this study, alanine aminotransferase or aspartate aminotransferase levels higher than 3 times the upper limit of normal associated with total bilirubin levels higher than 2 times the upper limit of normal were considered as serious AEs. Furthermore, any suspected transmission of an infectious agent via the Investigational Medicinal Product was also considered as an SAE.
Arm/Group | Inpatients | Outpatients
All-Cause Mortality (participants affected / at risk) | 1/136 | 0/38
Serious Adverse Events (participants affected / at risk) | 10/136 | 4/38
Other Adverse Events (participants affected / at risk) | 73/136 | 23/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inpatients (N=136) | Outpatients (N=38)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cholera (Infections and infestations) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 2 (2) | 1 (1)
Tuberculous pleurisy (Infections and infestations) | 1 (1) | 0 (0)
Uterine rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Starvation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0)
Psychomotor skills impaired (Nervous system disorders) | 1 (1) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Transverse presentation (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inpatients (N=136) | Outpatients (N=38)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 20 (24) | 7 (7)
Salivary hypersecretion (Gastrointestinal disorders) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 35 (41) | 6 (6)
Asthenia (General disorders) | 22 (24) | 1 (1)
Feeling hot (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 16 (16) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (1)
Dizziness (Nervous system disorders) | 10 (11) | 2 (2)
Headache (Nervous system disorders) | 24 (30) | 8 (8)
Tremor (Nervous system disorders) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 9 (10) | 3 (3)
Insomnia (Psychiatric disorders) | 12 (12) | 7 (7)
Hot flush (Vascular disorders) | 1 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
There is an overlap between the safety profile of fexinidazole and the g-HAT symptoms, making the interpretation of the safety data (in particular the relationship with fexinidazole) difficult as this was a cohort study and not a comparative study.

Some study sites were involved in another clinical trial. A recruitment bias towards patients not filling the other trial's criteria (pregnant and breastfeeding women, children, and patients with Karnofsky score between 40 and 50) may have occurred.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor authorizes publications by a single site provided that multicentric results are published beforehand and that any communication is submitted to sponsor for review at least 28 days ahead of the expected date of publication. The sponsor can submit comments for a period of 28 days. Upon sponsor request, any confidential information will have to be removed from the communication before publishing.

DOCUMENTS (2):
  • Study Protocol (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT03025789/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT03025789/SAP_001.pdf